CLINICAL TRIAL: NCT06128421
Title: Individual Nutrition Support in HBV-ACLF Patients at Nutrition Risk: a Randomized Controlled Trail
Brief Title: Individual Nutrition Support in HBV-ACLF Patients at Nutrition Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL17
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Malnutrition; Hepatitis B,Chronic; Acute-On-Chronic Liver Failure; Nutrition Support
MeSH Terms: conditions — Malnutrition; Hepatitis B, Chronic; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trail Group (Experimental): 30 patients will receive dietary counseling and individual nutrition support treatment based on Oral nutrition supplements and supplemented by parenteral nutrition.
  Interventions: Dietary Supplement: Individual nutritional support
- Control Group (No Intervention): 30 patients will receive standard care food provided by the hospital kitchen according to their ability and desire, standard care food provided by the hospital kitchen.

INTERVENTIONS:
Dietary Supplement: Individual nutritional support — Nutritional products and route（oral, parenteral）is possible to reach goals
  Arms: Trail Group

SUMMARY:
This study aims to investigate the safety and efficacy of individual nutrition support for treating hepatitis b virus(HBV) related acute-on-chronic liver failure patients at nutrition risk

DETAILED DESCRIPTION:
The aims of the randomized-controlled trial are to test the hypothesis that in medical inpatients with HBV related ACLF at risk for undernutrition defined by the nutritional risk score (NRS 2002), tailored nutritional therapy to reach nutritional targets based on individualized nutritional counseling is a effective strategy to prevent mortality, morbidity and functional decline.

Sixty patients with HBV related ACLF will be enrolled in this study. The participants are divided into trial Patients in the trail group will receive individualized nutritional therapy to reach nutritional targets (caloric, protein, others) based on a predefined nutritional strategy.In control patients, according to patients' appetite, standard hospital nutrition will be served. Nutritional therapy may be started in control patients, if any sort of swallowing disorders develops or if patients need to be prepared for operation. All patients will be re-assessed daily during the hospital stay for nutritional intake and nutritional therapy may be escalated within first 3days ( oral supplements, parenteral nutrition) if targets are not met (at least 75% of targets).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 60 years old;
2. Clinical diagnosis of chronic hepatitis b virus infection(positive hepatitis b surface antigen or positive hepatitis b virus DNA >0.5 year
3. serum total bilirubin level ≥12 mg/dl
4. prothrombin time international ratio ≥1.5
5. NRS≥ 3points
6. COSSH-ACLF IIs <8.4 points

Exclusion Criteria:

1. Other active liver disease;
2. Hepatocellular carcinoma or other malignancy, HIV, Chronic kidney disease(CKD), diabetes, thyroid disease, cardiopulmonary disease, neuromuscular diseases, serious psychiatric disease;
3. Acute cholecystitis, acute pancreatitis, biliary obstruction, short bowel syndrome, intestinal obstruction, inflammatory bowel disease;
4. Severe complications or other organ failure including sever infection, gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal failure(AGI III-IV);
5. Pregnancy, BMI<18.5 or BMI ≥28，organ transplantation, bed-ridden;
6. Unable to ingest oral nutrition, contraindication against parenteral nutrition
7. Admitted with enteral or parenteral nutrition in the last week
8. expected hospital length of stay<3 days，.expected residence in Guangdong Province length of live< 90 days

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival at 30 days | 30 days
Transplant free survival at 90 days | 90 days

SECONDARY OUTCOMES:
L3-SMI as a marker of muscle mass | 30 days, 90days
  Third lumbar skeletal muscle index(L3-SMI) by CT scan
Grip as markers of muscle strength | 30 days, 90days
  Grip
Short Physical Performance Battery (SPPB) as markers of physical performance | 30 days, 90 days
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests.
Improvement in quality of life | 30 days, 90days
  Improvement in quality of life measured with the EuroQol Group 5-Dimension Self-Report Questionnaire on admission and during follow up measured by patient interview
length of hospital stay | days in the hospital within index hospitalisation and within the 30 days of follow up measured by patient interview and medical chart review
  days in the hospital within index hospitalisation and within the 90 days of follow up measured by patient interview and medical chart review
Energy intake | 10 days
  Protein-calorie intake as assessed by serial 24-hour dietary recall
hepatic adverse outcomes | 10days,30 days, 90 days
  hepatic encephalopathy，esophageal variceal hemorrhage，etc
Combined safety endpoints in regard to side effects from nutritional therapy | measured at day 10 and 30
  Number of participants with side effects from nutritional support including
  (a) adverse gastrointestinal effects (diarrhea, nausea, vomiting, abdominal pain, abdominal distention) assessed by patient interview (yes/no) b) Complications due to center catheter for parenteral nutrition assessed by medical chart review (c) Refeeding syndrome assessed by chart review (d) Acute pancreatitis defined as 2 out of 3 criteria: abdominal pain, 3-fold increase in lipase or amylase, characteristic imaging findings assessed by chart review (e) Liver or gall bladder dysfunction assessed by chart review (f) Hyperglycemia (defined as glucose levels persistent levels >10mmol/l in patients without diabetes or well controlled diabetes) assessed by medical chart review

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Luo Q, Wang P, Wang L, Zheng X, Zhang Y, Xu W, Peng L. Efficacy and safety of individual nutrition support in patients with hepatitis B virus-related acute-on-chronic liver failure at nutrition risk: a study protocol for a randomised controlled clinical trial. BMJ Open. 2024 Dec 9;14(12):e088832. doi: 10.1136/bmjopen-2024-088832. PMID 39653573